CLINICAL TRIAL: NCT05284318
Title: Effect of Antibiotic Treatment Course on Clinical Outcome After Two-stage Revision of Prosthetic Joint Infection: A Prospective Cohort Study.
Brief Title: Prospective Cohort Study on Antibiotic Course and Efficacy After Two-stage Revision in PJI.
Acronym: PACER-PJI
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Fang, Deputy chief physician, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MRCTA ECFAH of FMU 2021404
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Periprosthetic Joint Infection; Anti-Bacterial Agents
Keywords: Periprosthetic joint infection; Second-stage revision; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Antibiotics treatment — After receiving intravenous antibiotics treatment for 2 weeks, and clinician determines whether to continue with any antibiotics.

SUMMARY:
This is a multicenter prospective cohort study in which patients were evaluated by inclusion and exclusion criteria before phase II revision surgery. Eligible patients will be included in this study after signing the informed consent form. After the second stage revision, according to the patient's symptoms and examination results, the attending physician used a reasonable antibiotic treatment scheme (including intravenous and oral medication). All patients voluntarily participated in the study and signed informed consent. During the treatment period, all prospective patients underwent clinical evaluation at the time points of 1, 3, 6, 12, 18 and 24 months after the start of antibiotic treatment after phase II revision. The infection control rate of patients was evaluated by follow-up at least 2 years after operation, so as to analyze the effect of antibiotic treatment course after two-stage revision of periprosthetic joint infection.

DETAILED DESCRIPTION:
Inclusion criteria：

1. A diagnosis of PJI was made according to MSIS criteria
2. Received spacer implantation and a full course of antibiotic treatment (at least 6 weeks), the patient was clinically determined to have infection control and underwent secondary joint revision.
3. Age ≥18 years old
4. The patient voluntarily participated in the study, and was physically and mentally tolerant to the treatment process and various tests of the study. He has signed an informed consent form and passed the examination of all the hospital ethics committees participating in the study.

Exclusion criteria：

1. Follow up data were not available;
2. The investigator judged that the patient no longer met the criteria of the study due to compliance problems.

Recruiting time：2021.10 -2023.10.31 Interventions Group：No Sample size：500 Study Population Description: Patients who underwent secondary replantation surgery for prosthetic joint infection at the First Affiliated Hospital of Fujian Medical University and other sub-centers were selected.

ELIGIBILITY:
Inclusion Criteria:

- 1. A diagnosis of PJI was made according to MSIS criteria. 2. Received spacer implantation and a full course of antibiotic treatment (at least 6 weeks), the patient was clinically determined to have infection control and underwent secondary joint revision.

3. Age ≥18 years old. 4. The patient voluntarily participated in the study, and was physically and mentally tolerant to the treatment process and various tests of the study. He has signed an informed consent form and passed the examination of all the hospital ethics committees participating in the study.

Exclusion Criteria:

* 1. Follow-up data not available. 2. Researchers judge that patients no longer meet the standards of the study due to compliance problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent secondary replantation surgery for prosthetic joint infection at the First Affiliated Hospital of Fujian Medical University and other sub-centers were selected.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clearance rate of infection | 31, December，2026
  Number of subjects with infection cleared/total number of subjects who completed follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zhang, Director, Study Director — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
Within six months after the trial complete